CLINICAL TRIAL: NCT07130084
Title: Virtual Reality in Elective Caesarean Births Study (VREC)- A Feasibility Study for a Virtual-reality Based Tool to Improve Patient Reported Outcomes Following Elective Caesarean Section.
Brief Title: Virtual Reality in Elective Caesarean Births Study (VREC)
Acronym: VREC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Royal United Hospitals Bath NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Rebecca Leslie, Consultant in Anaesthesia, Royal United Hospitals Bath NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 24/WA/0033
Record Dates: First submitted 2025-08-12; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Anxiety; Pregnancy; Pain
Keywords: Virtual reality
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality educational film (Experimental): The intervention arm will receive the standard antenatal care and pre-operative education plus will view the Virtual Reality Educational Film
  Interventions: Other: Virtual Reality Educational Film
- Control arm (No Intervention): The control arm will receive all standard antenatal care and pre-operative education

INTERVENTIONS:
Other: Virtual Reality Educational Film — The Virtual Reality Educational Film will be viewed during the antenatal appointment, post randomisation. The women will have access to the film at home should they want to watch it more than once.
  Arms: Virtual reality educational film

SUMMARY:
This study will establish the safety of a known intervention in a novel setting. It will assess how maternal anxiety during the peri-operative period of an elective cesarean section (eCS) is affected by the introduction of a virtual reality (VR) tool. A cesarean section is the most common operation performed in the world. Indeed, locally, we perform approximately 450 eCS annually, equating to 10% of all births. High maternal anxiety in the peri-operative period is well recognised. Although anxiety is considered to be an emotional response it has many physiological consequences which can confer significant morbidity. These include an increased pain perception (with higher analgesic requirement), increased length of hospital stay and a higher risk of infection. Providing high-quality pre-operative information to help patients reduce their anxiety has been used in other medical fields. The use of VR to deliver this information to paediatric populations has been shown to be particularly effective. VR has had limited scope outside of this population and we wish to change this.

Women booked for an eCS at the Royal United Hospital (RUH) will be eligible to participate. A bespoke VR tool (a video of a woman's journey through the process of an elective section at the RUH) will be shown to one group of women prior to eCS whilst another group will receive the standard preoperative information.

A series of quantitative and qualitative data points will be collected across both groups assessing their anxiety and satisfaction with the birthing process throughout the peri-operative period. The two groups will then be compared.

Recruitment will occur prior to the birth during scheduled appointments with the Midwifery team. If proven to be a safe intervention, we hope to run a larger study aiming to determine the efficacy and role of VR in improving maternal outcomes in cesarean births.

DETAILED DESCRIPTION:
The Royal College of Obstetrics and Gynaecology (RCOG) has a well-defined framework for involving pregnant women in research studies (clinical governance document 6a). They promote research in obstetrics but stress the key is that research should be completed 'with women, not on women'. For each step of the study, the RCOG framework will be adhered to.

Overview of the study and why it is important

An elective caesarean section (eCS) can be a very anxiety inducing time. Prior to the research project commencing, we developed a questionnaire that all women at Royal United Hospital, Bath (RUH) completed prior to their eCS. This demonstrated consistently high anxiety levels across obstetric populations, including those who had previous emergency caesarean sections. The main source of anxiety was often a fear 'of the unknown' and not knowing what to expect.

Although anxiety is considered to be an emotional response it has many physiological consequences which can confer significant morbidity. These include an increased pain perception (with higher analgesic requirement), increased length of hospital stay and a higher risk of post-operative wound infection.

The purpose of this study is to assess the safety of a virtual reality education film (VREF). The VR will provide a 360degree, 3-dimensional virtual tour demonstrating what will happen on their day of delivery, from entering Bath Birthing Centre through to being on the postnatal ward with their new baby. They will be able to watch this, if they choose, using a head set to make the experience more realistic. The ultimate purpose of the film is to reduce that fear of the unknown by giving patients and their families a detailed view of their upcoming journey.

Given the prevalence of high maternal anxiety and the potential emotional and physical costs of anxiety, it is important to try and develop new interventions to reduce this. However, the safety of any potential intervention is paramount. This study will assess the safety of our VREF.

Step 1: Creating the virtual reality video and writing the script RCOG states that service users should be involved in the development and delivery of the trial. We have already addressed this by involving patients via our PPI (patient and pubic involvement) where we have discussed with the women what they would like to see in the video, when and how they would like to view the video and how they would like the video to help them. We have incorporated all of this information into the script for our virtual reality education film (VREF). The script has been reviewed by multiple health professionals including midwives, obstetricians and anaesthetists to ensure a balanced and accurate view of an eCS is provided. It has also been read by patients prior to their eCS and their feedback has been taken into account for the final version of the script.

We have also discussed how the women feel about the VR element. The VR has been well received, with the main feedback being how useful it will be to be able to 'scroll' around the theatre/wards to fully orientate themselves prior to their eCS.

Step 2: Recruitment to study Potential participants will be identified and given information (patient information leaflet) about the study on an ad hoc basis when booked for their elective LSCS at any point during their pregnancy (as long as it's prior to 38 weeks gestation); this can be done by either their obstetrician or the research midwives.

Approved posters will be on the walls of the antenatal clinic with information about the study and contact details.

Research midwives will then contact the patients by phone to invite them for a formal appointment to consent at 38 weeks. Many patients will be attending hospital at around 38-39 weeks for obstetric follow up, so if feasible, research appointments will be aligned with this. If patients are not attending routinely, we will invite them for an appointment with the research midwives at an alternative time.

Formal consent will be sought at the appointment. Given that this study will only be undertaken for elective procedures, all patients will have plenty of time to weigh up the information provided to them before consenting to research and will be able to withdraw from the study any time.

RCOG states the importance of providing the service user with multiple ways to access information about the trial. Is also advises that any information leaflets should be produced in conjunction with the service user to ensure that they are easy to understand as well as accurate. The women will have access to both.

Step 3: Randomisation and baseline anxiety scores and cortisol levels Randomisation will be performed by a computer on a 1:1 basis to eliminate any bias. Patients that are randomised to the control arm will not have their care disadvantaged in any way. They will receive all the standard antenatal care and normal information that we provide prior to an eCS.

All women who consent to the study will require baseline scores for

* State Trait Anxiety Inventory Scale-5
* Visual Analogue Scale for Anxiety
* Serum Cortisol These will be carried out at the 38-39 week routine appointment at DAU to again reduce any additional trips to the hospital. The two anxiety scales/indexes are well validated having been used extensively in research projects across many populations and there are no ethical concerns regarding these.

A blood sample will need to taken for serum cortisol. The women always have a blood sample taken at this appointment to obtain a valid 'Group& Save' and Full Blood Count prior to surgery so there will be no additional venepuncture. All venepuncture and handling of blood products will be carried out by trained personnel in accordance with the Trust's guidelines and policies. For patients randomised to the intervention arm, they will be shown this video during their visit to DAU (Day Assessment Unit). As per the RCOG framework, the welfare of the woman and baby will take priority over any research, and the patients can stop watching the film at any time if they wish to do so.

After watching the VREF they will be able to ask the midwifery team any questions they might have. They will also be given access so they can watch the VREF on their own devices at home if they wish. The women in the intervention arm will also be provided with all the standard antenatal care and information to ensure they are not disadvantaged in any way.

Step 4: Day of elective caesarean section During the day of the eCS, the health and welfare of the woman and baby will be the absolute priority. We will ensure the women understand that they can withdraw from the study at any time during the day or in the recovery period and that this will not affect their care or treatment in any way.

During the day, there will be three time points at which we ask the patients to complete the following; On admission

* State Trait Anxiety Inventory Scale 5
* Visual Analogue Scale for Anxiety
* Serum Cortisol At skin closure
* State Trait Anxiety Inventory Scale 5
* Visual Analogue Scale for Anxiety
* Serum Cortisol 2 hours post-LSCS
* State Trait Anxiety Inventory Scale 5
* Visual Analogue Scale for Anxiety
* Serum Cortisol
* Patient satisfaction score
* Visual Analogue Scores for pain The serum cortisol level (blood test) will need to be taken at all three time points. Wherever possible this will be coordinated with the need for routine venepuncture/cannulation to reduce unnecessary venepuncture. Again, these samples will be taken by appropriately trained professionals to minimise the risk of repeated attempts.

Further information surrounding the birth such as time of birth, time of anaesthesia and fetal APGAR's will be collected unobtrusively by the anaesthetist to give the woman time to bond with her baby once delivered.

Step 5: Day after elective caesarean section

All women will remain an inpatient for at least 24 hours following a caesarean section so we will not need to women to re-attend hospital to gather any follow up data. The following data will be collected:

* Patient satisfaction score
* State Trait Anxiety Inventory Scale 5
* Visual Analogue Scale for Anxiety
* Visual Analogue Scores for pain
* Analgesia consumption in first 24 hours post-LSCS
* Time to breastfeed post-LSCS
* Time to mobilise post-LSCS This data will only be collected if the woman is happy to answer the questions, and we will ensure it is a convenient time for the mother to answer these questions. Again, keeping the welfare of the mother and baby at the forefront.

The following data will be collected from the patient's notes or anaesthetic chart (a sticker will be attached to the anaesthetic chart for the anaesthetist to complete):

* Time of anaesthesia
* Time of adequate block
* Time of birth
* Time of closing of the skin
* Did the mother have skin-to-skin with baby? What time?
* Fetal 5-minute APGAR
* Any unexpected events

Use of Virtual Reality in research

A brief literature review demonstrates there are at least 890 studies assessing virtual reality and anxiety. Virtual reality has been proven to be safe and accepted across multiple populations, including the paediatric population. A VR video was developed by J-H Ryu et al. for paediatric patients about to undergo an elective operation. The video gives them a tour of the operating suite prior to surgery. They report that it was well accepted by patients and their carers' and also demonstrated a reduction in pre-operative anxiety.

There is more limited use of VR in the obstetric population, but studies do exist. For example, Frey et al used VR during labour to assess its use as an analgesic. They again found VR to be an acceptable intervention and found it reduced both perceived pain and anxiety during labour.

In 'Health and safety implications of virtual reality: a review of empirical evidence' , Sharples and Patel discuss some of the potential health and safety implications. The main area they identify if the potential for nausea if fully immersive headsets are used. In our study, the use of headsets are fully optional, and women can stop using a headset at any time if it was causing any nausea.

Overall, virtual reality is a safe and well accepted intervention across multiple populations. We will carefully monitor for any adverse effects and stop the trial immediately if there were any concerns.

Inclusion/Exclusion Criteria:

Patients undergoing elective lower segment caesarean section (LSCS) at the Royal United Hospital, Bath.

Eligibility:

* Have had the decision for elective LSCS by 38 weeks gestation.
* Has never had an emergency or elective section previously
* Have a procedure planned and performed as a category 4 LSCS (an elective LSCS booked at a time that suits both the woman and obstetric team)
* Have use of an android or iOS operating system smartphone or tablet device.
* Have access to the internet.
* Have an active email address.
* Have capacity to consent to participate in the study.

Exclusion criteria:- Patient <18 years of age.- Patient refusal.- Women more likely to have atypical anxiety-related behaviour, restricted to:- Patients with a current severe mental health disorder under the care of the perinatal mental health team- Patients with medical or obstetric co-morbidities requiring pre-determined admission to maternity HDU care

* Congenital structural abnormalities requiring pre-determined admission to NICU- Patients where spinal anaesthesia is contra-indicated.- Patients who do not have access to a smart phone/computer

Withdrawal criteria

* Emergency LSCS - those in the following standardised categories of urgency as set out by NICE[23].

  * Category 1 - immediate threat to life of woman or fetus
  * Category 2 - maternal or fetal compromise which is not immediately life-threatening
  * Category 3 - no maternal or fetal compromise but needs early birth
* Women who receive a general anaesthetic.

Information Governance:

As per the RCOG guidelines, patient confidentiality will be maintained at all time. All data will be entered into a Trust based computer that is password protected. Subject names will be kept on a database and will be linked only with a study identification number for this research. There will be no patient identifiers. Only the research team will have access to this computer. Personal data will be stored in a locked office and maintained for 12 months after the completion of the study. Research data generated by the study will be stored for 5 years. Data will be collected and retained in accordance with the Data Protection Act 1998.

ELIGIBILITY:
Inclusion Criteria:

* Have had the decision for elective LSCS by 38 weeks gestation.
* Has never had an emergency or elective section previously
* Have a procedure planned and performed as a category 4 LSCS (an elective LSCS booked at a time that suits both the woman and obstetric team)
* Have use of an android or iOS operating system smartphone or tablet device.
* Have access to the internet.
* Have an active email address.
* Have capacity to consent to participate in the study.

Exclusion Criteria:

* Patient <18 years of age
* Patient refusal
* Patients who have had an emergency or elective LSCS previously.
* Patients with a history of anxiety disorders
* Patients with medical or obstetric co-morbidities requiring pre-determined admission to maternity HDU care
* Congenital structural abnormalities requiring pre-determined admission to NICU
* Patients where spinal anaesthesia is contra-indicated
* Women who have English of an insufficient standard to comprehend the consent and assessment process
* Prisoners

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10-14 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
patient feedback questionnaire after watching virtual reality education film | from enrollment up to 1 weeks post cesarean section
  Patients will complete a feedback questionnaire to assess if a pre-operative virtual reality education film is safe, feasible and acceptable intervention in women who have had an elective Cesarean section.

SECONDARY OUTCOMES:
State Trait Anxiety Inventory Scale 5 | from enrollment up to 48 hours post cesarean section
  The State-Trait Anxiety Inventory (STAI) is a commonly used measure of anxiety. It has 5 items for assessing anxiety. Each item is self rated on a score or 1-4 (1= not at all; 4=very much so). Item statements are: 'I feel upset', 'I feel frightened', 'I feel nervous', 'I feel jittery', and 'I feel confused'.
  STAI is completed at 5 time points (T1 at pre-clerking (approximately 38-39 weeks gestation), T2 on admission for LSCS, T3 at skin closure, T4 2 hour's post-LSCS, T5 at 24 hours post-LSCS patient will be phoned if they have left the hospital).
Visual Analogue Scale for Anxiety | from enrollment up to 48 hours post delivery
  VAS-A is a validated, self-reported instrument assessing anxiety. Participants are asked to indicate their level of anxiety on a scale from 0-10 (number 0 indicates no anxiety and the number 10 indicates severe anxiety)
  VAS-A at 5 time points (T1 at pre-clerking approximately 38-39 weeks gestation, T2 on admission for LSCS, T3 at skin closure, T4 2 hours post-LSCS, T5 at 24 hours post-LSCS patient will be phoned if they have left the hospital ) (Score 0-10).
Serum cortisol | From enrollment up to 48 hours post delivery
  Cortisol is a hormone and levels can alter depending on the stress response. It requires a blood test and will be measured at 4 time points (T1 at pre-clerking at approximately 38-39 weeks gestation, T2 on admission for LSCS, T3 at skin closure, T4 at 2 hours post-LSCS)
Patient satisfaction scores | enrollment up to 48 hours post cesarean section
  Participants are asked to rate their satisfaction on the care they received on a scale 0 -10, where 0 is very poor and 10 is extremely satisfied.
  Scores at two time points (T4 at 2 hours post-LSCS and T5 at 24 hours post-LSCS, patient will be phoned if they have left the hospital)(Score 0-10)
Visual Analogue Scores (VAS) for pain | up to 48 hours post cesarean section
  VAS-P is a validated, self-reported instrument for assessing pain in the peri-operative period. Participants are asked to select a point on the scale indicating the level of pain they are feeling. The number 0 indicates no pain and the number 10 indicates the worse pain possible
  This is performed at two time points (T4 at 2 hours post-LSCS, T5 at 24 hours post-LSCS patient will be phoned if they have left the hospital) (Score 0 to 10)
Analgesia consumption | from delivery up to 48hours post delivery
  Analgesia consumption in first 24 hours post-LSCS (amount of morphine in mg)

CONTACTS AND LOCATIONS:
Locations (1):
- Bath Birthing Centre, Royal United Hospital Bath Foundation Trust, Bath, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared. Only aggregated, anonymised results will be published.

REFERENCES:
- [Background] Zsido AN, Teleki SA, Csokasi K, Rozsa S, Bandi SA. Development of the short version of the spielberger state-trait anxiety inventory. Psychiatry Res. 2020 Sep;291:113223. doi: 10.1016/j.psychres.2020.113223. Epub 2020 Jun 12. PMID 32563747
- [Background] Kindler CH, Harms C, Amsler F, Ihde-Scholl T, Scheidegger D. The visual analog scale allows effective measurement of preoperative anxiety and detection of patients' anesthetic concerns. Anesth Analg. 2000 Mar;90(3):706-12. doi: 10.1097/00000539-200003000-00036. PMID 10702461
- [Background] Mackenzie JW. Daycase anaesthesia and anxiety. A study of anxiety profiles amongst patients attending a day bed unit. Anaesthesia. 1989 May;44(5):437-40. doi: 10.1111/j.1365-2044.1989.tb11349.x. PMID 2787129
- [Background] Jiang L, Zhang K, He W, Zhu X, Zhou P, Lu Y. Perceived Pain during Cataract Surgery with Topical Anesthesia: A Comparison between First-Eye and Second-Eye Surgery. J Ophthalmol. 2015;2015:383456. doi: 10.1155/2015/383456. Epub 2015 May 4. PMID 26064671
- [Background] North MM, North SM. Virtual reality therapy. In: Computer-assisted and web- based innovations in psychology, special education, and health. London: lsevier; 2016. p. 141-56.
- [Background] Dehghan F, Jalali R, Bashiri H. The effect of virtual reality technology on preoperative anxiety in children: a Solomon four-group randomized clinical trial. Perioper Med (Lond). 2019 Jun 4;8:5. doi: 10.1186/s13741-019-0116-0. eCollection 2019. PMID 31171963
- [Background] Sjoling M, Nordahl G, Olofsson N, Asplund K. The impact of preoperative information on state anxiety, postoperative pain and satisfaction with pain management. Patient Educ Couns. 2003 Oct;51(2):169-76. doi: 10.1016/s0738-3991(02)00191-x. PMID 14572947
- [Background] Gammon J, Mulholland CW. Effect of preparatory information prior to elective total hip replacement on psychological coping outcomes. J Adv Nurs. 1996 Aug;24(2):303-8. doi: 10.1046/j.1365-2648.1996.17911.x. PMID 8858434
- [Background] Johnston M, Vogele C. Benefits of psychological preparations for surgery: a meta-analysis. Annuals of Behavioural Medicine. 1993; 15: 245-56.
- [Background] Devine EC. Effects of psychoeducational care for adult surgical patients: a meta-analysis of 191 studies. Patient Educ Couns. 1992 Apr;19(2):129-42. doi: 10.1016/0738-3991(92)90193-m. PMID 1299818
- [Background] Hobson JA, Slade P, Wrench IJ, Power L. Preoperative anxiety and postoperative satisfaction in women undergoing elective caesarean section. Int J Obstet Anesth. 2006 Jan;15(1):18-23. doi: 10.1016/j.ijoa.2005.05.008. Epub 2005 Oct 26. PMID 16256338
- [Background] Gorkem U, Togrul C, Sahiner Y, Yazla E, Gungor T. Preoperative anxiety may increase postcesarean delivery pain and analgesic consumption. Minerva Anestesiol. 2016 Sep;82(9):974-80. Epub 2016 Mar 30. PMID 27028449
- [Background] Schupp CJ, Berbaum K, Berbaum M, Lang EV. Pain and anxiety during interventional radiologic procedures: effect of patients' state anxiety at baseline and modulation by nonpharmacologic analgesia adjuncts. J Vasc Interv Radiol. 2005 Dec;16(12):1585-92. doi: 10.1097/01.RVI.0000185418.82287.72. PMID 16371522
- [Background] Chieng YJ, Chan WC, Klainin-Yobas P, He HG. Perioperative anxiety and postoperative pain in children and adolescents undergoing elective surgical procedures: a quantitative systematic review. J Adv Nurs. 2014 Feb;70(2):243-55. doi: 10.1111/jan.12205. Epub 2013 Jul 19. PMID 23865442
- [Background] Carr E, Brockbank K, Allen S, Strike P. Patterns and frequency of anxiety in women undergoing gynaecological surgery. J Clin Nurs. 2006 Mar;15(3):341-52. doi: 10.1111/j.1365-2702.2006.01285.x. PMID 16466484
- [Background] Pokharel K, Bhattarai B, Tripathi M, Khatiwada S, Subedi A. Nepalese patients' anxiety and concerns before surgery. J Clin Anesth. 2011 Aug;23(5):372-8. doi: 10.1016/j.jclinane.2010.12.011. PMID 21802628
- [Background] Navarro-Garcia MA, Marin-Fernandez B, de Carlos-Alegre V, Martinez-Oroz A, Martorell-Gurucharri A, Ordonez-Ortigosa E, Prieto-Guembe P, Sorbet-Amostegui MR, Indurain-Fernandez S, Elizondo-Sotro A, Irigoyen-Aristorena MI, Garcia-Aizpun Y. [Preoperative mood disorders in patients undergoing cardiac surgery: risk factors and postoperative morbidity in the intensive care unit]. Rev Esp Cardiol. 2011 Nov;64(11):1005-10. doi: 10.1016/j.recesp.2011.06.009. Epub 2011 Sep 15. Spanish. PMID 21924811
- [Background] Caumo W, Ferreira MB. Perioperative anxiety: Psychobiology and effects in postoperative recovery. Pain Clin 2003;15:87 101.
- [Background] Hepp P, Hagenbeck C, Burghardt B, Jaeger B, Wolf OT, Fehm T, Schaal NK; MAGIC Group. Measuring the course of anxiety in women giving birth by caesarean section: a prospective study. BMC Pregnancy Childbirth. 2016 May 18;16:113. doi: 10.1186/s12884-016-0906-z. PMID 27188222
- [Background] Wyatt SS, Jones DA, Peach MJ, Gurrin L. Anxiety in patients having caesarean section under regional anaesthesia: a questionnaire and pilot study. Int J Obstet Anesth. 2001 Oct;10(4):278-83. doi: 10.1054/ijoa.2001.0866. PMID 15321585
- [Background] Speilberger CD Gorsuch RL, Lushene RE, Vagg P & Jacobs G. 1983. State-trait Anxiety Inventory (STAI). Mind garden, Menlo Park, CA.
- See also: 23. National Institute for Health and Care Excellence Clinical Excellence, (31st March 2021), Caesarean Birth [NICE guideline no. 192] — https://www.nice.org.uk/guidance/ng192/resources/caesarean-birth-pdf-66142078788805

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-13): https://cdn.clinicaltrials.gov/large-docs/84/NCT07130084/Prot_SAP_000.pdf